CLINICAL TRIAL: NCT05459181
Title: Molecular Outcome Surveillance Using AlloSure and AlloMap Guided Immunomodulation in Cardiac Transplant
Brief Title: HeartCare Immuno-optimization in Cardiac Allografts (MOSAIC)
Acronym: MOSAIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SN-C-00021
Record Dates: First submitted 2022-06-22; First posted 2022-07-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplant; Immunosuppression; Allograft
Keywords: HeartCare; Allograft loss and survival; Calcineurin inhibitors; Chronic immunosuppression; Steroid avoidance; Donor-specific antibodies; Donor-derived cell-free DNA; AlloSure; AlloMap; Gene expression profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control arm (No Intervention): 465 participants undergoing standard of care post-transplant surveillance
- Intervention arm (Experimental): 465 participants undergoing HeartCare protocol surveillance
  Interventions: Diagnostic Test: HeartCare

INTERVENTIONS:
Diagnostic Test: HeartCare — Using HeartCare platform as a tool to successfully augment immunosuppressant agents through regular surveillance allowing minimization of doses and number of agents.
  Arms: Intervention arm

SUMMARY:
This is an unblinded, randomized, controlled, two-arm interventional research study enrolling patients who are undergoing heart transplantation. The aim of the study is to determine whether patients at low risk of rejection can safely reduce the doses of their post-transplant immunosuppression medications using a combination of tests that include donor-specific antibodies (DSA), histology (looking at tissue from the donor heart), donor-derived cell-free DNA (AlloSure), and gene expression profiling (AlloMap). Eligible participants will be randomized in a 1:1 ratio into the HeartCare immune-optimization (intervention) arm or the corresponding observational (control) arm. AlloSure and AlloMap are the components of the HeartCare panel developed by CareDx.

DETAILED DESCRIPTION:
This is an open-label randomized controlled two-arm interventional trial. Eligible patients starting triple maintenance therapy (tacrolimus, mycophenolate mofetil and prednisone) post-transplant will be randomized at a 1:1 ratio into the HeartCare immuno-optimization (intervention) arm or the corresponding observational (control) arm. Participants enrolled in the study will begin HeartCare testing as specified in the protocol. All centers will use their own induction regimen provided that the induction practice represents standard of care. Participants will be randomized at 4-weeks post-transplant, assuming they meet requisite clinical/laboratory/histological criteria to proceed. In the Interventional Arm, participants will begin stepwise optimization of their immunosuppression regimen based on their HeartCare, clinical DSA testing, and histology. Patient data (including diagnosis and biopsy outcomes) will be collected through an electronic data capture portal where key results will be transcribed from the hospital EMR into the portal.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant recipients <2 weeks post-transplant
2. Patients aged 18 years or older
3. Planned post-transplant maintenance immunosuppression regimen consisting of prednisolone, tacrolimus and mycophenolate
4. Female participants of childbearing potential must be willing to ensure that they or their partner use effective contraception during the trial and for 3 months thereafter
5. Participant is willing and able to give informed consent for participation in the trial
6. In the Investigator's opinion, is able and willing to comply with all trial requirements

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

1. Multi-visceral transplant recipients
2. Female participant who is pregnant, lactating or planning pregnancy during the trial
3. Heart transplant recipients undergoing desensitization protocols prior to transplant based off high immunological risk profiles (determined by treating clinician)
4. Chronic oral steroid use for any reason that cannot be tapered off and discontinued
5. Planned post-transplant immunosuppression regimen utilizing cyclosporine, azathioprine, mTOR inhibitors, and/or co-stimulatory blockers
6. Contraindication to having AlloSure or AlloMap testing
7. Participant with life expectancy of less than 6 months or is inappropriate for immuno-optimization (including those patients at increased risk of primary disease recurrence w/ reduction in post-transplant immunosuppression)
8. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial. This includes clinical events that would significantly impact post-transplant immunosuppression such as major infectious complications or significant rejection episodes within the first month post-transplant.
9. Participants who are currently or have previously participated in another research trial involving an investigational immunological drug in the past 12 weeks
10. Any condition that would preclude protocol biopsies

Randomization Criteria (assessed at Week 4)

The participant may not proceed with randomization if ANY of the following apply at Week 4 post-transplant:

1. Maintenance immunosuppression that includes cyclosporine, azathioprine, mTOR inhibitors, and/or co-stimulatory blockers
2. Any episodes of biopsy-proven acute rejection (ACR ≥2R or AMR*)
3. Abnormal molecular profile defined as AlloSure >0.2%
4. Allograft dysfunction defined as LVEF <45%
5. eGFR <30mL/min
6. Presence of DSA (persistence of any pre-transplant DSA or dnDSA) *AMR 1 (H+) with DSA/graft dysfunction or AMR > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Allograft loss at 12-months post-transplant (safety) | 12 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Incidence of Allograft loss at 24-months post-transplant (safety) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Total number of acute rejection episodes (ACR >2R or AMR*) at 12-months post-transplant (safety) | 12 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Total number of acute rejection episodes (ACR >2R or AMR*) at 24-months post-transplant (safety) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
EQ-5D survey performed at 12-months post-transplant to assess allograft function (safety) | 12 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
TTE imaging performed at 12-months post-transplant to assess allograft function (safety) | 12 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
EQ-5D survey performed at 24-months post-transplant to assess allograft function (safety) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
TTE imaging performed at 24-months post-transplant to assess allograft function (safety) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Incidence of dnDSA formation at 12-months post-transplant (safety and efficacy) | 12 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Incidence of dnDSA formation at 24-months post-transplant (safety and efficacy) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Change in eGFR at 12-months post-transplant (efficacy) | 12 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Change in eGFR at 24-months post-transplant (efficacy) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.
Total number of biopsies performed post-transplant, including both surveillance and clinically indicated biopsies (efficacy) | 24 months
  Demonstrate the safety and efficacy of HeartCare as a tool to successfully optimize immunosuppressant agents using regular surveillance for safe drug minimization.

SECONDARY OUTCOMES:
Histological assessment of tissue biopsy with paired AlloSure dd-cfDNA and AlloMap GEP results (HeartCare) - performed both 'For Cause' and 'Surveillance' using standard biopsy assessment. | 6 months
  Identify correlation between HeartCare and histopathological allograft rejection based on all clinical biopsies.
Association between AlloSure dd-cfDNA and AlloMap GEP (HeartCare) results with successful immuno-optimization, longitudinal clinical/laboratory parameters (dnDSA), and histologic data (allograft rejection, CAV). | 24 months
  Establish temporal relationships between HeartCare and allograft injury patterns such as dnDSA formation, allograft rejection and CAV.
Data collection from patient medical record, to capture episodes of infection, viral PCR results, changes in immunosuppression and treatment of rejection, as well as all adverse advents. | 24 months
  Assessment of all medical events throughout the duration of the study.